CLINICAL TRIAL: NCT06940609
Title: Magnetic Resonance Analysis of Neural Inflammatory Factors and External Stimulation (MANIFEST)
Brief Title: Magnetic Resonance Analysis of Neural Inflammatory Factors and External Stimulation
Acronym: MANIFEST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: The Mind Research Network (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 24-470; HT9425-24-1-0742 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-04-02; First posted 2025-04-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Long COVID; Long COVID Syndrome; Long COVID-19 Syndrome; PASC; PASC Post Acute Sequelae of COVID 19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham accelerated iTBS (Sham Comparator): Sham stimulation is delivered using the same coil as active stimulation, producing an equivalent sound, however it is shielded so that no effective magnetic field reaches the participant's brain. To blind participants to active versus sham condition, a mild electrical skin stimulation that has no brain effects is delivered simultaneously with iTBS at the scalp to both active and sham groups, creating the same sense of skin sensation in both groups.
  Interventions: Device: accelerated intermittent theta burst stimulation
- Active accelerated iTBS (Experimental): Participants will be assigned to receive fMRI-guided iTBS (5 days, 5 sessions/day) to the left dorsolateral prefrontal cortex (dlPFC) during the sham-controlled phase. Each participant is invited to undergo 25 more sessions (5 more days) of open label, unblinded active accelerated fMRI-guided iTBS to the left dlPFC.
  Interventions: Device: accelerated intermittent theta burst stimulation

INTERVENTIONS:
Device: accelerated intermittent theta burst stimulation — Intermittent theta burst stimulation (iTBS), a FDA-approved form of noninvasive neuromodulation, can reduce neuropsychiatric symptoms and modulate inflammation in the thalamus as detected using dMRS, suggesting a potentially effective and efficient treatment approach with a pathophysiological component that is readily quantifiable.

SUMMARY:
The goal of this clinical trial is to test whether a type of rapid outpatient brain stimulation that uses magnetic fields, called accelerated intermittent theta burst stimulation (iTBS), can treat symptoms such as brain fog, depression, and anxiety in patients with Long COVID. The main questions it aims to answer are:

* Is iTBS effective and feasible for reducing Long COVID symptoms? We will measure these symptoms using the Symptom Burden Questionnaire.
* Are there changes in inflammatory brain chemicals associated with treatment with iTBS? We will be looking at levels of choline in the brain, which is thought to be related to inflammation.

Researchers will compare sham versus active forms of iTBS to see if the active group has greater improvement in symptoms.

Participants will complete symptom surveys, cognitive tests, and magnetic resonance imaging scans at the beginning, middle, and end of treatment.

DETAILED DESCRIPTION:
Chronic neuropsychiatric symptoms of post-acute sequelae of COVID-19 (neuro-PASC) can lead to disability, loss of function, and reduced quality of life, but there are currently no validated effective treatments. We propose a randomized sham-controlled trial of "Magnetic Resonance Analysis of Neural Inflammatory Factors and External Stimulation (MANIFEST)." We will deliver active or sham accelerated iTBS (5x/day, 10 days, 25 blinded sessions followed by 25 open-label sessions) to each participant's brain target. We will assess neuro-PASC symptoms, mood, anxiety, cognition, and quality of life from baseline to end-of-treatment. We will correlate symptom improvement with clinical and imaging variables.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-80
2. a documented diagnosis of PASC with evidence of ongoing symptoms as demonstrated by score of 12 on the NIH RECOVER Symptom List
3. have "brain fog" or cognitive difficulties as one of the ongoing symptoms
4. are fluent in English
5. if taking psychotropic medications, have been on stable doses for the past month.

Exclusion Criteria:

1. a prior history of other neurological disease, or any history of seizures, so as to reduce risk of exacerbation of epilepsy or other neurological symptoms;
2. history of a psychotic disorder, such as schizophrenia or bipolar disorder, so as to reduce risk of psychiatric decompensation
3. history of ongoing substance/alcohol dependence, to reduce confounding effects on diagnosis and brain imaging
4. presence of any implanted electrical device (e.g., pacemaker), to reduce risk of device malfunction from rTMS
5. recent medical hospitalization (within four weeks), to reduce risk of medical decompensation during the study
6. any condition that would prevent the subject from completing the protocol
7. appointment of a legal representative, to avoid coercion of a vulnerable population
8. any ongoing litigation related to medical diagnosis, or disability, to prevent interference with legal proceedings
9. any contraindication to MRI
10. membership in an identified vulnerable population, including minors, pregnant women, and prisoners, so as to prevent coercion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Aim 1 | From baseline to end of treatment at 2 weeks
  Demonstrate that accelerated iTBS is effective and feasible for reducing neuro-PASC symptoms. Change in the score in the "Cognitive Function/Brain Fog Symptoms" score from the PACS: Post-acute COVID-19 Syndrome Questionnaire, where low scores are more severe symptoms compared to higher scores. Scale 1-Severly Unable to 4-Able. Higher scores show improvement in symptoms.
Aim 2 | From baseline to end of treatment at 2 weeks
  Identify neurometabolic and structural features associated with outcomes in MANIFEST. ADCcho in the thalamus measured using dMRS. The apparent diffusion coefficient of choline (ADCcho) is a measure of activity of microglia, higher values indicate higher levels of microglia. Decreased ADCcho means less microglia activation, and less inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Davin Quinn, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Science Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographics, symptoms, cognitive testing, and imaging data.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Genovese G, Marjanska M, Auerbach EJ, Cherif LY, Ronen I, Lehericy S, Branzoli F. In vivo diffusion-weighted MRS using semi-LASER in the human brain at 3 T: Methodological aspects and clinical feasibility. NMR Biomed. 2021 May;34(5):e4206. doi: 10.1002/nbm.4206. Epub 2020 Jan 13. PMID 31930768
- [Background] Schubert J, Tonietto M, Turkheimer F, Zanotti-Fregonara P, Veronese M. Supervised clustering for TSPO PET imaging. Eur J Nucl Med Mol Imaging. 2021 Dec;49(1):257-268. doi: 10.1007/s00259-021-05309-z. Epub 2021 Mar 29. PMID 33779770
- [Background] Ling JM, Klimaj S, Toulouse T, Mayer AR. A prospective study of gray matter abnormalities in mild traumatic brain injury. Neurology. 2013 Dec 10;81(24):2121-7. doi: 10.1212/01.wnl.0000437302.36064.b1. Epub 2013 Nov 20. PMID 24259552
- [Background] Mayer AR, Hanlon FM, Dodd AB, Ling JM, Klimaj SD, Meier TB. A functional magnetic resonance imaging study of cognitive control and neurosensory deficits in mild traumatic brain injury. Hum Brain Mapp. 2015 Nov;36(11):4394-406. doi: 10.1002/hbm.22930. Epub 2015 Aug 19. PMID 26493161
- [Background] Mayer AR, Yang Z, Yeo RA, Pena A, Ling JM, Mannell MV, Stippler M, Mojtahed K. A functional MRI study of multimodal selective attention following mild traumatic brain injury. Brain Imaging Behav. 2012 Jun;6(2):343-54. doi: 10.1007/s11682-012-9178-z. PMID 22673802
- [Background] Mayer AR, Toulouse T, Klimaj S, Ling JM, Pena A, Bellgowan PS. Investigating the properties of the hemodynamic response function after mild traumatic brain injury. J Neurotrauma. 2014 Jan 15;31(2):189-97. doi: 10.1089/neu.2013.3069. Epub 2013 Nov 20. PMID 23965000
- [Background] Davenport ND, Lim KO, Armstrong MT, Sponheim SR. Diffuse and spatially variable white matter disruptions are associated with blast-related mild traumatic brain injury. Neuroimage. 2012 Feb 1;59(3):2017-24. doi: 10.1016/j.neuroimage.2011.10.050. Epub 2011 Oct 20. PMID 22040736
- [Background] Davenport ND, Lamberty GJ, Nelson NW, Lim KO, Armstrong MT, Sponheim SR. PTSD confounds detection of compromised cerebral white matter integrity in military veterans reporting a history of mild traumatic brain injury. Brain Inj. 2016;30(12):1491-1500. doi: 10.1080/02699052.2016.1219057. PMID 27834537
- [Background] Meier TB, Bellgowan PS, Singh R, Kuplicki R, Polanski DW, Mayer AR. Recovery of cerebral blood flow following sports-related concussion. JAMA Neurol. 2015 May;72(5):530-8. doi: 10.1001/jamaneurol.2014.4778. PMID 25730545
- [Background] Mayer AR, Stephenson DD, Wertz CJ, Dodd AB, Shaff NA, Ling JM, Park G, Oglesbee SJ, Wasserott BC, Meier TB, Witkiewitz K, Campbell RA, Yeo RA, Phillips JP, Quinn DK, Pottenger A. Proactive inhibition deficits with normal perfusion after pediatric mild traumatic brain injury. Hum Brain Mapp. 2019 Dec 15;40(18):5370-5381. doi: 10.1002/hbm.24778. Epub 2019 Aug 28. PMID 31456319
- [Background] Katz I, Barry CN, Cooper SA, Kasprow WJ, Hoff RA. Use of the Columbia-Suicide Severity Rating Scale (C-SSRS) in a large sample of Veterans receiving mental health services in the Veterans Health Administration. Suicide Life Threat Behav. 2020 Feb;50(1):111-121. doi: 10.1111/sltb.12584. Epub 2019 Aug 23. PMID 31441952
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Hughes SE, Haroon S, Subramanian A, McMullan C, Aiyegbusi OL, Turner GM, Jackson L, Davies EH, Frost C, McNamara G, Price G, Matthews K, Camaradou J, Ormerod J, Walker A, Calvert MJ. Development and validation of the symptom burden questionnaire for long covid (SBQ-LC): Rasch analysis. BMJ. 2022 Apr 27;377:e070230. doi: 10.1136/bmj-2022-070230. PMID 35477524
- [Background] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062
- [Background] Sasaki N, Yamatoku M, Tsuchida T, Sato H, Yamaguchi K. Effect of Repetitive Transcranial Magnetic Stimulation on Long Coronavirus Disease 2019 with Fatigue and Cognitive Dysfunction. Prog Rehabil Med. 2023 Feb 28;8:20230004. doi: 10.2490/prm.20230004. eCollection 2023. PMID 36861061
- [Background] Noda Y, Sato A, Shichi M, Sato A, Fujii K, Iwasa M, Nagano Y, Kitahata R, Osawa R. Real world research on transcranial magnetic stimulation treatment strategies for neuropsychiatric symptoms with long-COVID in Japan. Asian J Psychiatr. 2023 Mar;81:103438. doi: 10.1016/j.ajp.2022.103438. Epub 2022 Dec 28. PMID 36610206
- [Background] Chang CH, Chen SJ, Chen YC, Tsai HC. A 30-Year-Old Woman with an 8-Week History of Anxiety, Depression, Insomnia, and Mild Cognitive Impairment Following COVID-19 Who Responded to Accelerated Bilateral Theta-Burst Transcranial Magnetic Stimulation Over the Prefrontal Cortex. Am J Case Rep. 2023 Apr 2;24:e938732. doi: 10.12659/AJCR.938732. PMID 37004143
- [Background] Nakatomi Y, Mizuno K, Ishii A, Wada Y, Tanaka M, Tazawa S, Onoe K, Fukuda S, Kawabe J, Takahashi K, Kataoka Y, Shiomi S, Yamaguti K, Inaba M, Kuratsune H, Watanabe Y. Neuroinflammation in Patients with Chronic Fatigue Syndrome/Myalgic Encephalomyelitis: An (1)(1)C-(R)-PK11195 PET Study. J Nucl Med. 2014 Jun;55(6):945-50. doi: 10.2967/jnumed.113.131045. Epub 2014 Mar 24. PMID 24665088
- [Background] Qanneta R. Long COVID-19 and myalgic encephalomyelitis/chronic fatigue syndrome: Similarities and differences of two peas in a pod. Reumatol Clin (Engl Ed). 2022 Dec;18(10):626-628. doi: 10.1016/j.reumae.2022.05.001. No abstract available. PMID 36435560
- [Background] Salari N, Khodayari Y, Hosseinian-Far A, Zarei H, Rasoulpoor S, Akbari H, Mohammadi M. Global prevalence of chronic fatigue syndrome among long COVID-19 patients: A systematic review and meta-analysis. Biopsychosoc Med. 2022 Oct 23;16(1):21. doi: 10.1186/s13030-022-00250-5. PMID 36274177
- [Background] Luo J, Feng Y, Li M, Yin M, Qin F, Hu X. Repetitive Transcranial Magnetic Stimulation Improves Neurological Function and Promotes the Anti-inflammatory Polarization of Microglia in Ischemic Rats. Front Cell Neurosci. 2022 Apr 12;16:878345. doi: 10.3389/fncel.2022.878345. eCollection 2022. PMID 35496902
- [Background] Sun P, Fang L, Zhang J, Liu Y, Wang G, Qi R. Repetitive Transcranial Magnetic Stimulation for Patients with Fibromyalgia: A Systematic Review with Meta-Analysis. Pain Med. 2022 Mar 2;23(3):499-514. doi: 10.1093/pm/pnab276. PMID 34542624
- [Background] Chen X, Yin L, An Y, Yan H, Zhang T, Lu X, Yan J. Effects of repetitive transcranial magnetic stimulation in multiple sclerosis: A systematic review and meta-analysis. Mult Scler Relat Disord. 2022 Mar;59:103564. doi: 10.1016/j.msard.2022.103564. Epub 2022 Jan 29. PMID 35123289
- [Background] Aftanas LI, Gevorgyan MM, Zhanaeva SY, Dzemidovich SS, Kulikova KI, Al'perina EL, Danilenko KV, Idova GV. Therapeutic Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Neuroinflammation and Neuroplasticity in Patients with Parkinson's Disease: a Placebo-Controlled Study. Bull Exp Biol Med. 2018 Jun;165(2):195-199. doi: 10.1007/s10517-018-4128-4. Epub 2018 Jun 19. PMID 29923005
- [Background] Chou PH, Lu MK, Tsai CH, Hsieh WT, Lai HC, Shityakov S, Su KP. Antidepressant efficacy and immune effects of bilateral theta burst stimulation monotherapy in major depression: A randomized, double-blind, sham-controlled study. Brain Behav Immun. 2020 Aug;88:144-150. doi: 10.1016/j.bbi.2020.06.024. Epub 2020 Jun 24. PMID 32592861
- [Background] Zhao X, Li Y, Tian Q, Zhu B, Zhao Z. Repetitive transcranial magnetic stimulation increases serum brain-derived neurotrophic factor and decreases interleukin-1beta and tumor necrosis factor-alpha in elderly patients with refractory depression. J Int Med Res. 2019 May;47(5):1848-1855. doi: 10.1177/0300060518817417. Epub 2019 Jan 7. PMID 30616482
- [Background] Chen J, Zeng Y, Hong J, Li C, Zhang X, Wen H. Effects of HF-rTMS on microglial polarization and white matter integrity in rats with poststroke cognitive impairment. Behav Brain Res. 2023 Feb 15;439:114242. doi: 10.1016/j.bbr.2022.114242. Epub 2022 Nov 28. PMID 36455674
- [Background] Zuo C, Cao H, Feng F, Li G, Huang Y, Zhu L, Gu Z, Yang Y, Chen J, Jiang Y, Wang F. Repetitive transcranial magnetic stimulation exerts anti-inflammatory effects via modulating glial activation in mice with chronic unpredictable mild stress-induced depression. Int Immunopharmacol. 2022 Aug;109:108788. doi: 10.1016/j.intimp.2022.108788. Epub 2022 Apr 30. PMID 35504201
- [Background] Sasso V, Bisicchia E, Latini L, Ghiglieri V, Cacace F, Carola V, Molinari M, Viscomi MT. Repetitive transcranial magnetic stimulation reduces remote apoptotic cell death and inflammation after focal brain injury. J Neuroinflammation. 2016 Jun 14;13(1):150. doi: 10.1186/s12974-016-0616-5. PMID 27301743
- [Background] Stekic A, Zeljkovic M, Zaric Kontic M, Mihajlovic K, Adzic M, Stevanovic I, Ninkovic M, Grkovic I, Ilic TV, Nedeljkovic N, Dragic M. Intermittent Theta Burst Stimulation Ameliorates Cognitive Deficit and Attenuates Neuroinflammation via PI3K/Akt/mTOR Signaling Pathway in Alzheimer's-Like Disease Model. Front Aging Neurosci. 2022 May 17;14:889983. doi: 10.3389/fnagi.2022.889983. eCollection 2022. PMID 35656538
- [Background] Tian L, Sun SS, Cui LB, Wang SQ, Peng ZW, Tan QR, Hou WG, Cai M. Repetitive Transcranial Magnetic Stimulation Elicits Antidepressant- and Anxiolytic-like Effect via Nuclear Factor-E2-related Factor 2-mediated Anti-inflammation Mechanism in Rats. Neuroscience. 2020 Mar 1;429:119-133. doi: 10.1016/j.neuroscience.2019.12.025. Epub 2020 Jan 7. PMID 31918011
- [Background] Clarke D, Beros J, Bates KA, Harvey AR, Tang AD, Rodger J. Low intensity repetitive magnetic stimulation reduces expression of genes related to inflammation and calcium signalling in cultured mouse cortical astrocytes. Brain Stimul. 2021 Jan-Feb;14(1):183-191. doi: 10.1016/j.brs.2020.12.007. Epub 2020 Dec 24. PMID 33359601
- [Background] Medina-Fernandez FJ, Escribano BM, Padilla-Del-Campo C, Drucker-Colin R, Pascual-Leone A, Tunez I. Transcranial magnetic stimulation as an antioxidant. Free Radic Res. 2018 Apr;52(4):381-389. doi: 10.1080/10715762.2018.1434313. Epub 2018 Mar 2. PMID 29385851
- [Background] Guo B, Zhang M, Hao W, Wang Y, Zhang T, Liu C. Neuroinflammation mechanisms of neuromodulation therapies for anxiety and depression. Transl Psychiatry. 2023 Jan 9;13(1):5. doi: 10.1038/s41398-022-02297-y. PMID 36624089
- [Background] Rawlinson C, Jenkins S, Thei L, Dallas ML, Chen R. Post-Ischaemic Immunological Response in the Brain: Targeting Microglia in Ischaemic Stroke Therapy. Brain Sci. 2020 Mar 11;10(3):159. doi: 10.3390/brainsci10030159. PMID 32168831
- [Background] Urenjak J, Williams SR, Gadian DG, Noble M. Proton nuclear magnetic resonance spectroscopy unambiguously identifies different neural cell types. J Neurosci. 1993 Mar;13(3):981-9. doi: 10.1523/JNEUROSCI.13-03-00981.1993. PMID 8441018
- [Background] Reischauer C, Gutzeit A, Neuwirth C, Fuchs A, Sartoretti-Schefer S, Weber M, Czell D. In-vivo evaluation of neuronal and glial changes in amyotrophic lateral sclerosis with diffusion tensor spectroscopy. Neuroimage Clin. 2018;20:993-1000. doi: 10.1016/j.nicl.2018.10.001. Epub 2018 Oct 3. PMID 30317156
- [Background] Ercan E, Magro-Checa C, Valabregue R, Branzoli F, Wood ET, Steup-Beekman GM, Webb AG, Huizinga TW, van Buchem MA, Ronen I. Glial and axonal changes in systemic lupus erythematosus measured with diffusion of intracellular metabolites. Brain. 2016 May;139(Pt 5):1447-57. doi: 10.1093/brain/aww031. Epub 2016 Mar 11. PMID 26969685
- [Background] Genovese G, Palombo M, Santin MD, Valette J, Ligneul C, Aigrot MS, Abdoulkader N, Langui D, Millecamps A, Baron-Van Evercooren A, Stankoff B, Lehericy S, Petiet A, Branzoli F. Inflammation-driven glial alterations in the cuprizone mouse model probed with diffusion-weighted magnetic resonance spectroscopy at 11.7 T. NMR Biomed. 2021 Apr;34(4):e4480. doi: 10.1002/nbm.4480. Epub 2021 Jan 21. PMID 33480101
- [Background] Kappelmann N, Dantzer R, Khandaker GM. Interleukin-6 as potential mediator of long-term neuropsychiatric symptoms of COVID-19. Psychoneuroendocrinology. 2021 Sep;131:105295. doi: 10.1016/j.psyneuen.2021.105295. Epub 2021 Jun 3. PMID 34119855
- [Background] Salvio G, Gianfelice C, Firmani F, Lunetti S, Balercia G, Giacchetti G. Bone Metabolism in SARS-CoV-2 Disease: Possible Osteoimmunology and Gender Implications. Clin Rev Bone Miner Metab. 2020;18(4):51-57. doi: 10.1007/s12018-020-09274-3. Epub 2020 Sep 1. PMID 32904892
- [Background] Gentile S, Strollo F, Mambro A, Ceriello A. COVID-19, ketoacidosis and new-onset diabetes: Are there possible cause and effect relationships among them? Diabetes Obes Metab. 2020 Dec;22(12):2507-2508. doi: 10.1111/dom.14170. Epub 2020 Aug 27. No abstract available. PMID 32790021
- [Background] Peleg Y, Kudose S, D'Agati V, Siddall E, Ahmad S, Nickolas T, Kisselev S, Gharavi A, Canetta P. Acute Kidney Injury Due to Collapsing Glomerulopathy Following COVID-19 Infection. Kidney Int Rep. 2020 Apr 28;5(6):940-945. doi: 10.1016/j.ekir.2020.04.017. eCollection 2020 Jun. No abstract available. PMID 32346659
- [Background] Muccioli L, Pensato U, Cani I, Guarino M, Cortelli P, Bisulli F. COVID-19-Associated Encephalopathy and Cytokine-Mediated Neuroinflammation. Ann Neurol. 2020 Oct;88(4):860-861. doi: 10.1002/ana.25855. Epub 2020 Aug 14. No abstract available. PMID 32715524
- [Background] Mehandru S, Merad M. Pathological sequelae of long-haul COVID. Nat Immunol. 2022 Feb;23(2):194-202. doi: 10.1038/s41590-021-01104-y. Epub 2022 Feb 1. PMID 35105985
- [Background] Schultheiss C, Willscher E, Paschold L, Gottschick C, Klee B, Henkes SS, Bosurgi L, Dutzmann J, Sedding D, Frese T, Girndt M, Holl JI, Gekle M, Mikolajczyk R, Binder M. The IL-1beta, IL-6, and TNF cytokine triad is associated with post-acute sequelae of COVID-19. Cell Rep Med. 2022 Jun 21;3(6):100663. doi: 10.1016/j.xcrm.2022.100663. PMID 35732153
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Cabaro S, D'Esposito V, Di Matola T, Sale S, Cennamo M, Terracciano D, Parisi V, Oriente F, Portella G, Beguinot F, Atripaldi L, Sansone M, Formisano P. Cytokine signature and COVID-19 prediction models in the two waves of pandemics. Sci Rep. 2021 Oct 21;11(1):20793. doi: 10.1038/s41598-021-00190-0. PMID 34675240
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Del Valle DM, Kim-Schulze S, Huang HH, Beckmann ND, Nirenberg S, Wang B, Lavin Y, Swartz TH, Madduri D, Stock A, Marron TU, Xie H, Patel M, Tuballes K, Van Oekelen O, Rahman A, Kovatch P, Aberg JA, Schadt E, Jagannath S, Mazumdar M, Charney AW, Firpo-Betancourt A, Mendu DR, Jhang J, Reich D, Sigel K, Cordon-Cardo C, Feldmann M, Parekh S, Merad M, Gnjatic S. An inflammatory cytokine signature predicts COVID-19 severity and survival. Nat Med. 2020 Oct;26(10):1636-1643. doi: 10.1038/s41591-020-1051-9. Epub 2020 Aug 24. PMID 32839624
- [Background] Boldrini M, Canoll PD, Klein RS. How COVID-19 Affects the Brain. JAMA Psychiatry. 2021 Jun 1;78(6):682-683. doi: 10.1001/jamapsychiatry.2021.0500. No abstract available. PMID 33769431
- [Background] Proal AD, VanElzakker MB. Long COVID or Post-acute Sequelae of COVID-19 (PASC): An Overview of Biological Factors That May Contribute to Persistent Symptoms. Front Microbiol. 2021 Jun 23;12:698169. doi: 10.3389/fmicb.2021.698169. eCollection 2021. PMID 34248921
- [Background] Graham EL, Clark JR, Orban ZS, Lim PH, Szymanski AL, Taylor C, DiBiase RM, Jia DT, Balabanov R, Ho SU, Batra A, Liotta EM, Koralnik IJ. Persistent neurologic symptoms and cognitive dysfunction in non-hospitalized Covid-19 "long haulers". Ann Clin Transl Neurol. 2021 May;8(5):1073-1085. doi: 10.1002/acn3.51350. Epub 2021 Mar 30. PMID 33755344
- [Background] Ronen I, Ercan E, Webb A. Axonal and glial microstructural information obtained with diffusion-weighted magnetic resonance spectroscopy at 7T. Front Integr Neurosci. 2013 Mar 13;7:13. doi: 10.3389/fnint.2013.00013. eCollection 2013. PMID 23493316
- [Background] De Marco R, Ronen I, Branzoli F, Amato ML, Asllani I, Colasanti A, Harrison NA, Cercignani M. Diffusion-weighted MR spectroscopy (DW-MRS) is sensitive to LPS-induced changes in human glial morphometry: A preliminary study. Brain Behav Immun. 2022 Jan;99:256-265. doi: 10.1016/j.bbi.2021.10.005. Epub 2021 Oct 18. PMID 34673176
- [Background] Sherif ZA, Gomez CR, Connors TJ, Henrich TJ, Reeves WB; RECOVER Mechanistic Pathway Task Force. Pathogenic mechanisms of post-acute sequelae of SARS-CoV-2 infection (PASC). Elife. 2023 Mar 22;12:e86002. doi: 10.7554/eLife.86002. PMID 36947108
- [Background] Badenoch JB, Rengasamy ER, Watson C, Jansen K, Chakraborty S, Sundaram RD, Hafeez D, Burchill E, Saini A, Thomas L, Cross B, Hunt CK, Conti I, Ralovska S, Hussain Z, Butler M, Pollak TA, Koychev I, Michael BD, Holling H, Nicholson TR, Rogers JP, Rooney AG. Persistent neuropsychiatric symptoms after COVID-19: a systematic review and meta-analysis. Brain Commun. 2021 Dec 17;4(1):fcab297. doi: 10.1093/braincomms/fcab297. eCollection 2022. PMID 35169700
- [Background] Sonneville R, Dangayach NS, Newcombe V. Neurological complications of critically ill COVID-19 patients. Curr Opin Crit Care. 2023 Apr 1;29(2):61-67. doi: 10.1097/MCC.0000000000001029. PMID 36880556
- [Background] Chen C, Haupert SR, Zimmermann L, Shi X, Fritsche LG, Mukherjee B. Global Prevalence of Post-Coronavirus Disease 2019 (COVID-19) Condition or Long COVID: A Meta-Analysis and Systematic Review. J Infect Dis. 2022 Nov 1;226(9):1593-1607. doi: 10.1093/infdis/jiac136. PMID 35429399
- [Background] Xie Y, Bowe B, Al-Aly Z. Burdens of post-acute sequelae of COVID-19 by severity of acute infection, demographics and health status. Nat Commun. 2021 Nov 12;12(1):6571. doi: 10.1038/s41467-021-26513-3. PMID 34772922
- [Background] Richard SA, Pollett SD, Lanteri CA, Millar EV, Fries AC, Maves RC, Utz GC, Lalani T, Smith A, Mody RM, Ganesan A, Colombo RE, Colombo CJ, Lindholm DA, Madar C, Chi S, Huprikar N, Larson DT, Bazan SE, English C, Parmelee E, Mende K, Laing ED, Broder CC, Blair PW, Chenoweth JG, Simons MP, Tribble DR, Agan BK, Burgess TH; EPICC COVID-19 Cohort Study Group. COVID-19 Outcomes Among US Military Health System Beneficiaries Include Complications Across Multiple Organ Systems and Substantial Functional Impairment. Open Forum Infect Dis. 2021 Nov 10;8(12):ofab556. doi: 10.1093/ofid/ofab556. eCollection 2021 Dec. PMID 34909439